CLINICAL TRIAL: NCT01835821
Title: A Clinical Evaluation of Hand-veneered, Porcelain-fused NobelProcera(TM) Crown Shaded Zirconia and NobelProcera(TM) Full Contour Crown IPS e.Max CAD on Molars
Brief Title: Clinical Study of Porcelain-fused and IPS e.Max CAD Crowns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Prof. Marco Ferrari, Professor, University of Siena
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T-158; T-158s (Registry Identifier: T-158s)
Record Dates: First submitted 2013-04-05; First posted 2013-04-19 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Success; Survival; CDA Index
Keywords: zirconia; crown; IPS e.max CAD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- prosthesis (Experimental): NobelProcera™ Crown shaded zirconia:
  The device is an individual, ceramic core (figure a) made of shaded zirconium with an anatomic contour providing homogenous veneering material thickness and a minimum core thickness of 0.4 or 0.7mm. The core is veneered with dental porcelain (IPS e.max Ceram) at the dental laboratory
  Interventions: Device: prosthetic crowns

INTERVENTIONS:
Device: prosthetic crowns — prosthetic crowns

SUMMARY:
This clinical study has the objective to compare the longevity and the clinical behaviour (CDA Index, soft tissue behavior, success and survival rates) of single cemented ceramic crowns made with shaded zirconia (NobelProceraTM Shaded Zirconia) and NobelProceraTM full contour crowns IPS e.max CAD lithium disilicate on molars.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be at least 18 (or age of consent) and less than 70 at the time of inclusion.
* The subject is healthy and compliant with good oral hygiene.
* The subject is in need of at least two paired contalateral single-tooth full coverage molar restorations in the maxilla and/or mandible.
* The subject shall have a stable occlusal relationship with a fully restored, fixed opposing dentition.
* Obtained informed consent from the subject.
* No apical disorder or inflammation of abutment teeth, adjacent and opposing teeth.
* Good gingival / periodontal / periapical status of restoring, opposing and adjacent teeth. Healed situation of soft tissue augmentation is allowed.
* The subject is available for the 5-year term of the investigation.

Exclusion Criteria:

* The subject is not able to give her/his informed consent to participate.
* Alcohol or drug abuse as noted in patient records or in patient history.
* Reason to believe that the treatment might have a negative effect on the patient's total situation (psychiatric problems), as noted in patient records or in patient history.
* An existing condition where acceptable retention of the restoration is impossible to attain
* Mobility of the tooth to be restored.
* Pathologic pocket formation of 4 mm or greater around the tooth to be restored.
* Severe bruxism or other destructive habits.
* Amount of attached soft tissue is insufficient (no attached gingiva on the buccal side of the tooth).
* Health conditions, which do not permit the restorative procedure.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2010-03; Primary Completion 2015-09 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
success of Porcelain-fused and IPS e.Max CAD Crowns | 5 years
  A "successful crown" is when the CDA index (Marginal integrity, Color match, Surface texture and Anatomic form) shall be Romeo or Sierra (excellent or acceptable) at delivery and remain so during the study period.

SECONDARY OUTCOMES:
survival of Porcelain-fused and IPS e.Max CAD Crowns | 5 years
  A "surviving crown" is when the crown remains in occlusion, and when the subject's treatment is functionally successful even though all the individual success criteria are not fulfilled.

OTHER OUTCOMES:
CDA index | 5 years
  California Dental Association. Quality Evaluation for Dental Care. Guidelines for the Assessment of Clinical Quality and Professional Performance. Los Angeles: CDA, 1977.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dental Materials and Fixed Prosthodontics of Siena, Tuscan School of Dental Medicine, University of Florence and Siena, Siena, Italy, Siena, SI, Italy

REFERENCES:
- [Derived] Cagidiaco EF, Grandini S, Goracci C, Joda T. A pilot trial on lithium disilicate partial crowns using a novel prosthodontic functional index for teeth (FIT). BMC Oral Health. 2019 Dec 9;19(1):276. doi: 10.1186/s12903-019-0957-4. PMID 31818278